CLINICAL TRIAL: NCT00832832
Title: Eyelid Closure in Topical Glaucoma Therapy
Brief Title: Eyelid Closure in Glaucoma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Henry D. Jampel, M.D., M.H.S., Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00021272
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; Eye drop; Intraocular pressure; Eyelid closure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eyelid closure (Experimental): Eyelids will be closed after administration of eye drop
  Interventions: Other: Eyelid closure
- No eyelid closure (Active Comparator): Eyelids will not be closed after eye drop instillation
  Interventions: Other: No intervention will be assigned

INTERVENTIONS:
Other: Eyelid closure — Eyelid will be closed after eye drop instillation
  Arms: Eyelid closure
Other: No intervention will be assigned — No intervention will be assigned to this arm
  Other Names: No intervention needed in Arm 2
  Arms: No eyelid closure

SUMMARY:
This research is being done to determine if closing your eyelids after you take your glaucoma drops makes them more effective in lowering your eye pressure, and to determine if closing your eyelids for 5 minutes is better than closing them for one minute

DETAILED DESCRIPTION:
* Abstract

  * Eye drops to lower intraocular pressure (IOP) remain the principal therapy for glaucoma. The path from the writing of a prescription of IOP-lowering drops to optimal lowering of IOP and preventing the development or worsening of glaucoma has many steps. One critical step is to maximize the amount of drug in the eye drop that reaches the target tissue in the eye once the eye drop is on the ocular surface. The literature supports the conclusion that eyelid closure (EC) and/or nasolacrimal occlusion (NLO) can increase the effect on IOP, decrease the frequency of dosing, and decrease blood levels. They do so by increasing the contact time of the applied drug with the ocular surface, and by decreasing the amount of drug that passes through the nasolacrimal duct and into the nasopharynx.
  * Fifteen years ago landmark studies were performed with pilocarpine and timolol. In retrospect, the principal limitations of these studies were that they empirically studied only one duration (5 minutes) of EC or NLO, and did not include (because they hadn't yet been invented) what are now the most commonly used eye drops to lower IOP, the prostaglandins. The limitation of the 5 minute duration is that it may be impractical for many patients and decrease adherence due to its inconvenience.
  * My research hypothesis is that EC used in conjunction with prostaglandin eye drop administration will result in greater IOP lowering and that 1 minute of EC may be as effective as 5 minutes.
  * The research is potentially of great clinical importance. Pharmaceutical companies invest heavily in developing and marketing eye drops that may be 1 mm Hg more effective than their competitors. If similar or greater improvements can be made with a simple patient action, patient care will be improved
* Objectives (include all primary and secondary objectives)

  * To determine if EC increases the IOP lowering effect of prostaglandin eye drops.
  * To determine the relative effectiveness of EC of 1 and 5 minute duration.
* Study Procedures

  * Controlled clinical trial, using one eye of each subject as the experimental eye (EC plus drug) and the other as a control (drug alone). Half of the patients will perform EC for 1 minute; the other half for 5 minutes.
  * Subjects will be recruited from the glaucoma practices at Johns Hopkins Hospital and Wilmer at Greenspring Station. Eligibility (see 5 below) will be assessed during their regularly scheduled visit. Participants will sign consent forms and will be scheduled for 3 study visits, none of which will be part of routine clinical care. The subject will be instructed NOT to use his/her prostaglandin eye drop on the day preceding study visit 1.
  * Study visit 1-day 1 The subject will be instructed by the study coordinator in eyelid closure. The IOP will be measured 3 times in one 5 minute period between 7:30 and 10 am using Goldmann applanation tonometry and the median IOP will be recorded (baseline IOP). The subject will be randomized to performing eyelid closure in the right or left eye for either 1 or 5 minutes. Based on the randomization, the study coordinator will instill one drop of the prostaglandin eye drop (latanoprost, travoprost, or bimatoprost) that the patient normally uses into the appropriate eye, and observe the subject perform eyelid closure in the chosen eye for either 1 or 5 minutes.

One hour later, the IOP will be measured 3 times by an individual masked to which eye had EC and the median IOP will be recorded (1 hour IOP). The patient will be instructed NOT to use his/her prostaglandin eye drop that night and an appointment for the following morning will be scheduled.

* Study visit 2-day 2 The IOP will be measured 3 times in one 5 minute period between 7:30 and 10 am using Goldmann applanation tonometry by an individual masked to which eye had EC, and the median IOP will be recorded (24 hour IOP). The subject will be instructed to resume his/her prostaglandin that evening and will be instructed to continue EC at home in the selected eye for the designated amount of time (1 or 5 minutes) until the third study visit.
* Study visit 3-between day 8 and 15 The IOP will be measured 3 times between 7:30 and 10 am using Goldmann applanation tonometry, by an individual masked to which eye had EC, and the median IOP will be recorded (1 week IOP).

  * Study duration and number of study visits required of research participants.
* The total duration of the study is 1-2 weeks
* Blinding, including justification for blinding or not blinding the trial, if applicable.
* Subjects will not be masked. Masking of the IOP measurer is essential for avoiding bias
* Justification of why participants will not receive routine care or will have current therapy stopped.
* Subjects will be continuing their routine care throughout the study.
* Justification for inclusion of a placebo or non-treatment group.
* There is no placebo group.
* Definition of treatment failure or participant removal criteria.
* Participants will be removed if they are unable to perform EC or if they desire to leave the study
* Description of what happens to participants receiving therapy when study ends or if a participant's participation in the study ends prematurely.
* All subjects will be continuing the therapy that they were already taking before entering the study

  * Inclusion/Exclusion Criteria
* Inclusion - Patient must be using one of the three topical prostaglandins (latanop rost, travaprost, or bimatoprost), and no other IOP lowering eye drops for at least one month.
* Exclusion -Previous laser or incisional surgery for glaucoma. Use of punctual plugs Abnormal slit lamp exam (except for cataract or intraocular lens implant). No incisional eye surgery for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years, use of one of the three topical prostaglandins (latanoprost, travaprost, or bimatoprost), and no other IOP-lowering eye drops for at least one month.

Exclusion Criteria:

* Previous laser or incisional surgery for glaucoma, use of punctual plugs, an abnormal slit lamp exam (except for cataract or intraocular lens implant) and incisional eye surgery within the last 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Amount of intraocular pressure lowering | 24 hours

SECONDARY OUTCOMES:
Amount of intraocular pressure lowering | 1 hour and one week

CONTACTS AND LOCATIONS:
Overall Officials: Henry D Jampel, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins - The Wilmer Eye Institute, Baltimore, Maryland, United States